CLINICAL TRIAL: NCT02462018
Title: Effects of Functional Electrical Stimulation on Gait in Children With Hemiplegic and Diplegic Cerebral Palsy
Brief Title: Effects of Functional Electrical Stimulation on Gait in Children With Cerebral Palsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLV-0192-15
Record Dates: First submitted 2015-05-31; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-04

CONDITIONS: Cerebral Palsy, Congenital; Muscle Spasticity
Keywords: Cerebral Palsy; Muscle Spasticity; Orthoses; Functional Electrical Stimulation; Prospective
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WalkAide (Experimental)
  Interventions: Device: WalkAide

INTERVENTIONS:
Device: WalkAide — Patiants with hemiplegic or asymmetric diplegic CP will use WalkAide device for 4 months .First month for adjustment and three months of daily using of the device.
  For each patient two assessments will be conducted: at baseline and at post-intervention follow-up.
  During the assessments each child will go through:
  A. Medical interview and neurological and physical therapist examination. B. Motor function tests: "6 min walk test", Gross motor function measure (GMFM) ,"Timed up and down stairs test" (TUDS), walking on a ramp ,with and without the FES device.
  C. Gait analysis test with and without FES device. D. Parents will be requested to complete questionnaires on the frequency of falling.
  E. On the second assessment parents wiil be requested to complete a questionnaire about the compliance to the FES.

SUMMARY:
Cerebral palsy (CP) is the most common neuromuscular disorder among children, resulting from a non-progressive injury during early brain development which leads to impairment of movement and posture.

Muscle weakness and spasticity associated with CP limit the joint range of motion and negatively impact ambulatory ability. Most ambulatory children with CP are prescribed with ankle-foot orthoses (AFOs) to improve ankle position and stability and to maintain muscle range. Nevertheless, AFOs may also restrict desired motions and may exacerbate muscle weakness and atrophy.

During the last years a novel method is being used for treating upper motor neuron drop foot, by means of dynamic orthoses, namely Functional Electrical Stimulation (FES).

These FES devices cause dorsiflexion of foot by stimulating the peroneal nerve and activating the tibialis anterior muscle. Most of the studies of FES devices were conducted on adult population. These studies showed improvement in laboratory and functional gait parameters. There are relatively few studies on children with hemiplegic or diplegic CP with favorable results. There is no solid evidence whether the improvements seen in laboratory setting of children with CP, are reflected on functional ambulation in daily life. In addition, there are no defined parameters which could predict the response to FES among those children.

The aim of this study is to determine whether using FES device (WalkAide; Innovative Neurotronics, Austin, TX, USA) improves daily motor function and gait parameters in children with spastic hemiplegic or diplegic CP. additionally, we aim to define clinical and biomechanical parameters that can predict a favorable response to using the FES device.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common neuromuscular disorder among children, resulting from a non-progressive injury during early brain development which leads to impairment of movement and posture.

Individuals with CP exhibit a wide range of motor disabilities; however, approximately 70% of them achieve the ability to ambulate during childhood, albeit with difficulty.

Muscle weakness and spasticity associated with CP limit the joint range of motion and negatively impact ambulatory ability. The ankle joint is affected in virtually all patients. Insufficient ankle dorsiflexion during swing, foot drop and excessive plantar flexion during early to mid-stance may cause standing and walking instability with greater risk for falling. Most ambulatory children with CP are prescribed with ankle-foot orthoses (AFOs) to improve ankle position and stability for standing and walking and to maintain muscle range. Nevertheless, AFOs may also restrict desired motions and may exacerbate muscle weakness and atrophy, leading to further loss of function over time. In addition many children, especially adolescents, avoid using AFOs because of discomfort and concerns regarding negative effects on body image.

During the last years a novel method is being used for treating upper motor neuron drop foot, by means of dynamic orthoses, namely Functional Electrical Stimulation (FES).

These FES devices cause dorsiflexion of foot by stimulating the peroneal nerve and activating the tibialis anterior muscle.

FES devices, by actively stimulating the muscle have theoretical advantages over static AFOs. In addition the stimulator can be cosmetically better accepted.

Most of the studies of FES devices were conducted on adult population with upper motor neuron defect. These studies showed improvement in laboratory and functional gait parameters.In addition to the direct orthotic effect of the device during utilization, some studies also indicated a therapeutic effect ("carry over effect"), which was postulated to arise through the neural plasticity facilitation by increasing the strength of afferent feedback inputs to CNS. Whether this therapeutic effect actually exists and for how long is still unclear.

A variety of Functional Electrical Stimulation (FES) devices are being increasingly prescribed as a treatment option in CP children. There are relatively few studies on children with hemiplegic or diplegic CP. Prosser et al(Prosser et al 2013), reported good acceptability of FES device in CP population. Other studies have showed as well favorable results, with improvement of ankle kinematics parameters, such as dorsiflexion angle at swing phase and initial contact. Damiano et al (Damiano et al 2012) showed evidence of use-dependent muscle plasticity with increased tibialis anterior muscle thickness while using FES devices in CP patients.

There is still no solid evidence whether the improvements seen in laboratory setting are reflected on functional ambulation in daily life. Some studies showed improvement in walking speed while others did not.

Moreover, some studies also indicated an effect variability among subjects, which could be partially explained by the heterogeneity of CP population. There are no defined parameters which could predict the response to FES among those children.

The WalkAide(WalkAide; Innovative Neurotronics, Austin, TX, USA) is a battery-operated, small medical electrical stimulator device, which attaches to a molded cuff located just below the knee and produces controlled dorsiflexion of the foot during walk.It utilizes a tilt sensor and accelerometer to control the timing and duration of the stimulation during walking.Use of the Tilt Sensor to trigger stimulation eliminates the need for additional components or external wires.

The aim of this study is to determine whether using WalkAide device, improves daily motor function and gait parameters in children with spastic hemiplegic or diplegic CP. In addition, we aim to define clinical and biomechanical parameters that can predict a favorable response to using the FES device.

ELIGIBILITY:
Inclusion Criteria:

-Children above age of 6 years, with hemiplegic and asymmetric diplegic CP GMFCS I/II, with drop foot and dynamic contracture of the ankle on examination, who are being treated at the CP clinic at Tel Aviv Sourasky Medical Center, Tel Aviv, Israel.

Exclusion Criteria:

* Children with fixed contracture of ankle joint (passive range of motion< 0 degree); children who had orthopedic surgery to the leg or had botulinum toxin injection to the plantar or dorsiflexor muscles within the 6 months prior to the study; children who cannot tolerate the electrical stimulation delivered by the device.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
"Six min walk test" | 4 months
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (Maher C et al ,2008)
"Gross motor function measure" (GMFM) section E | 4 months
  The Gross Motor Function Measure (GMFM) is a clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. Section E evaluate walking, running and jumping skills (Rosenbaum PL et al, 2008)
"Timed up and down stairs test" | 4 months
  This test measures time going up and down 14-step flight of stairs (Zaino CA et al 2004)
Ankle angle at initial contact | 4 months
  measured by "Gait analysis laboratory"
Peak dorsiflexion angle in swing phase | 4 months
  measured by "Gait analysis laboratory"

REFERENCES:
- [Background] Prosser LA, Curatalo LA, Alter KE, Damiano DL. Acceptability and potential effectiveness of a foot drop stimulator in children and adolescents with cerebral palsy. Dev Med Child Neurol. 2012 Nov;54(11):1044-9. doi: 10.1111/j.1469-8749.2012.04401.x. Epub 2012 Aug 27. PMID 22924431
- [Background] LIBERSON WT, HOLMQUEST HJ, SCOT D, DOW M. Functional electrotherapy: stimulation of the peroneal nerve synchronized with the swing phase of the gait of hemiplegic patients. Arch Phys Med Rehabil. 1961 Feb;42:101-5. No abstract available. PMID 13761879
- [Background] Maher CA, Williams MT, Olds TS. The six-minute walk test for children with cerebral palsy. Int J Rehabil Res. 2008 Jun;31(2):185-8. doi: 10.1097/MRR.0b013e32830150f9. PMID 18467936
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Zaino CA, Marchese VG, Westcott SL. Timed up and down stairs test: preliminary reliability and validity of a new measure of functional mobility. Pediatr Phys Ther. 2004 Summer;16(2):90-8. doi: 10.1097/01.PEP.0000127564.08922.6A. PMID 17057533